CLINICAL TRIAL: NCT01729234
Title: Effects of Dietary Nitrate Supplementation on Age-related Vascular Dysfunction
Brief Title: Effects of Dietary Nitrate on Age-related Vascular Function
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Nitrate for vascular age
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Endothelial Dysfunction
Keywords: age related Endothelial Dysfunction
MeSH Terms: interventions — Nitrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrate (Experimental): 150µmol /Kg bodyweight /day
  Interventions: Dietary Supplement: Nitrate
- PLacebo (Placebo Comparator): 150µmol /Kg bodyweight /day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nitrate — Dietary Supplement
  Arms: Nitrate
Dietary Supplement: Placebo — Dietary Supplement
  Arms: PLacebo

SUMMARY:
Purpose of the study is to characterize the chronic effect of dietary nitrate on vascular function in healthy volunteers with particular emphasis on age-related alterations.

ELIGIBILITY:
Inclusion Criteria:

>55 Years Healthy

Exclusion Criteria:

known cardiovascular disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Endothelial function measured by flow-mediated dilation (FMD) | 30 days
  The effect of dietary nitrate on endothelial function as measured by flow-mediated dilation (FMD) after forearm ischemia and reperfusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Heinrich-Heine-University, Düsseldorf, North Rhine-Westphalia, Germany